CLINICAL TRIAL: NCT06639100
Title: Real World Data and Patient Reported Outcomes in Diabetes: a Standard Set for Person-Centred Care in Emilia-Romagna During and After Covid-19
Brief Title: This Will Be an Observational, Exploratory Study Targeting a Population of Subjects with Diabetes from 4 Different Geographical Areas of Emilia- Romagna.
Acronym: REWINDER
Status: Active, not recruiting | Type: Observational
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Other Study IDs: REWINDER
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This will be an observational, exploratory study targeting a population of subjects with diabetes from 4 different geographical areas of Emilia- Romagna.

DETAILED DESCRIPTION:
Diabetes is a pivot condition involving a range of complications and interventions from multiple care providers over a long period of time. For this reason, it represents a critical field of chronic care where person-centred models can be better implemented using real world data on a continuous basis to support research and clinical practice. These activities are extremely challenging to carry out at national level, due to the lack of standardised definitions and clear guidelines on privacy and data protection, data exchange and statistical processing. We propose to implement a Regional Surveillance System for person-centred care in Diabetes that will be sustainable, standardised, actionable, introducing a value-based approach, privacy enhanced, statistically fair (internationally comparable), and clinically transparent, whose performance outputs will be made publicly available. This will be an observational, exploratory study targeting a population of subjects with diabetes from 4 different geographical areas of Emilia- Romagna. The study population will be followed up by 4 participating centres for 612 months, which already collect demographics, anthropometric data and clinical records at the Diabetes Outpatient Clinics using the same electronic format and data management software (Smart Digital Clinic from Meteda). Measurements for the target population will be available on a rolling basis, as they will be recorded as a part of routine care during ordinary visits. Further information will be acquired using other administrative sources, through data linkage of available databases: hospital discharge records, pharmaceutical prescriptions in and out of hospital, specialist visits, payment exemption and the primary master index (mortality records).The project will enroll all patients from 4 operational units (Romagna, Ferrara, Reggio Emilia and Parma). The UO "Diabetology" at "Azienda USL della Romagna" has a capacity of a total patient pool of 28,000 consecutive patients per year. The UO "Diabetology" at Azienda USL Reggio Emilia has a capacity of a total patient pool of 40,000 consecutive patients per year. The UO "Endocrinologia e Malattie del Metabolismo" at Azienda Ospedaliero- Universitaria Parma has a capacity of a total patient pool of 2,500 consecutive patients per year. The UO "Diabetology" at Azienda USL Ferrara has a capacity of a total patient pool of 5,000 consecutive patients per year. All centres collect personal data, anthropometric and clinical records of the Diabetes Outpatient Clinic using the same electronic format and data management software (Smart Digital Clinic from Meteda). Therefore, measurements for the target population will be available on a continuous basis, as they will be recorded as a part of routine care during ordinary visits.

This basis will be used to select 1,600 consecutive patients that will be followed up expanding the range of items available through a specific activity of data collection in the areas of PROMs and Covid-19. Each operating unit will recruit 400 patients (~100 with type 1 diabetes and ~300 with type 2 diabetes).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be all those recorded in 4 operational units with an "active status", defined as those who attended a visit during the last three years or booked one in the course of the study.

Participants will have T1D for at least 1 year and be aged ≥18 to <40 years. Patients with type 2 diabetes will have diabetes for at least 1 year. PROMs will be measured among subjects aged ≥40 to <70 years only.

Exclusion Criteria:

* Patients who deceased or migrated during the last three years prior to the start of the study.

Furthermore, we will exclude pregnant women, patients with known and recorded cognitive deficiency (eg, Down's syndrome, Alzheimer), severe somatic comorbidity (eg, end-stage renal disease, severe heart failure, severe cancer), and/or a major psychiatric diagnosis (eg, severe depression or bipolar disorder, schizophrenia) as diabetes distress is often neither ethical nor possible to discuss with these groups of patients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total population of 63,500 people with diabetes in 4 geographical areas of Emilia-Romagna.
Sampling Method: Probability Sample
Enrollment: 63500 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2024-10-26 (Estimated)

PRIMARY OUTCOMES:
PROMs | 12 mouth
  The primary outcome measure will be pre-post change in the 3 PROMs that will be measured in the study population.
  All items will be condensed for the whole population into observations at baseline (time 0) and, 6 months and one year. Patient reported outcomes (PROMs) will be collected at baseline and after 6 12 months. All data will be linked to the administrative records to build an all-embracing file, which, after anonymization of the data, will be used for statistical analysis. A specific study questionnaire including all questions for the validated PROMs will be filled at the clinical site, with the direct support of a specialised care providers. The questionnaire will be administered twice, at baseline and follow-up visit (after 6 12 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Ausl della Romagna Direttore UO di Diabetologia, Ravenna, RA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carinci F, Messina R, Michelini M, Bici A, Berardo A, Dei Cas A, Iezzi E, Di Iorio CT, Gualdi S, Aldigeri R, Fantini MP, Bonadonna RC, Massi Benedetti M, Di Bartolo P. Real-world data and patient-reported outcomes in diabetes in Emilia-Romagna (REWINDER): protocol of a federated cohort study for the regional evaluation of quality of care during and after COVID-19. BMJ Open. 2025 Oct 23;15(10):e102401. doi: 10.1136/bmjopen-2025-102401. PMID 41130696